CLINICAL TRIAL: NCT05157165
Title: Convalescent Plasma in Hospitalized COVID-19 Patients: a Single Center Experience
Brief Title: Convalescent Plasma in Hospitalized COVID-19 Patients
Status: No longer available | Type: Expanded Access
Sponsor: Azienda Socio Sanitaria Territoriale di Mantova (Other)
Responsible Party: Principal Investigator, Massimo Franchini, Director Immunohematology and Transfusion Center, Azienda Socio Sanitaria Territoriale di Mantova
Other Study IDs: 00001
Record Dates: First submitted 2021-12-10; First posted 2021-12-14 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

INTERVENTIONS:
Biological: Convalescent plasma — Hyperimmune plasma from convalescent COVID-19 donors with titre 1:80 or more

SUMMARY:
The study assesses the efficacy and safety of administration of hyperimmune plasma in hospitalized COVID-19 patients. Efficacy was measured as 28-day mortality following convalescent plasma transfusion. Safety was measured as the rate of adverse reactions. to plasma infusion.

DETAILED DESCRIPTION:
Inclusion criteria:

Adult inpatients with a severe form of COVID-19 have been enrolled, with at least one of the following inclusion criteria: 1) tachypnea with respiratory rate (RR) > 30 breaths/min; 2) oxygen saturation (SpO2) ≤ 93% at rest and in room air; 3) partial pressure of oxygen (PaO2)/fraction of inspired oxygen (FiO2) ≤ 200 mmHg, 4) radiological picture and/or chest CT scan showing signs of interstitial disease and/or rapid progression of lung involvement.

Primary outcome:

Overall mortality at 28 days after hospitalization

Secondary outcome:

Adverse reaction to plasma transfusion.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients admitted for severe COVID-19

Exclusion Criteria:

* < 18 years
* participation in any other clinical trial of an experimental treatment for COVID-19

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult